CLINICAL TRIAL: NCT02901613
Title: Prophylactic Post-Cesarean Incisional Negative-pressure Wound Therapy in Morbidly Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Peter R Cole, MD, Chief of Gynecology, Albany Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AlbanyMC1
Record Dates: First submitted 2016-09-11; First posted 2016-09-15 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Negative-pressure Wound Therapy; Morbid Obesity; Cesarean Section; Wound Infection
MeSH Terms: conditions — Obesity, Morbid; Wound Infection | interventions — Negative-Pressure Wound Therapy

ARMS (2):
- Retrospective (No Intervention): Standard dry sterile dressing
- Prospective (Experimental): Negative-pressure wound therapy
  Interventions: Device: Negative-pressure wound therapy

INTERVENTIONS:
Device: Negative-pressure wound therapy
  Arms: Prospective

SUMMARY:
To evaluate the effectiveness of negative-pressure wound therapy in decreasing wound complications in morbidly obese patients (BMI greater than of equal to 40) at Albany Medical Center Hospital. Retrospective data will be collected regarding morbidly obese patients who have undergone cesarean section and patients will be recruited to have the intervention (negative-pressure wound therapy) applied and outcomes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing cesarean section at Albany Medical Center Hospital
* Current BMI greater than or equal to 40

Exclusion Criteria:

* Current BMI less than 40
* current skin or soft tissue infection
* skin or soft tissue disorder
* allergy to silver

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Wound complication | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Cole, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States